CLINICAL TRIAL: NCT00399568
Title: Phase 3 Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Parallel, Multiple-Dose Study of the Analgesic Efficacy and Safety of IV Acetaminophen (APAP) Versus Placebo Over 48 Hours(Hrs) for the Treatment of Postoperative Pain After Gynecologic Surgery
Brief Title: Efficacy and Safety of Intravenous Acetaminophen Over 48 Hrs for the Treatment of Post-op Pain After Gynecologic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPI-APA-301
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Results first posted 2010-12-10 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-09

CONDITIONS: Postoperative Pain; Hysterectomy
Keywords: Pain; Gynecologic; IV Acetaminophen; Postoperative; Analgesic
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Acetaminophen; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV acetaminophen 1 g/100 mL solution (Experimental)
  Interventions: Drug: IV Acetaminophen
- IV Placebo 100 mL solution (Placebo Comparator)
  Interventions: Drug: IV Placebo 100 mL solution

INTERVENTIONS:
Drug: IV Acetaminophen — Intravenous acetaminophen 1 g/100 mL
  Other Names: IV Acetaminophen (IV APAP)
  Arms: IV acetaminophen 1 g/100 mL solution
Drug: IV Placebo 100 mL solution — IV Placebo 100 mL solution dosed at same frequency as IV Acetaminophen every 6 hours (q6h)
  Other Names: IV Placebo (non-active product)
  Arms: IV Placebo 100 mL solution

SUMMARY:
This study will be investigating the efficacy and safety administration of multiple doses of intravenous (IV) acetaminophen (IVAPAP) in the 48 hour period following Gynecologic Surgery.

DETAILED DESCRIPTION:
The research hypothesis is that IV Acetaminophen will provide greater reduction in pain intensity and greater pain relief for moderate and severe pain as compared to placebo in the 48 hours following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergo gynecologic surgery using standard abdominal approach such as midline or Pfannenstiel incision
* 18-75 years of age
* Body Mass Index (BMI) between 19-45
* American Society of Anesthesiologists (ASA) risk class of I, II, III
* Not have received neuraxial (spinal or epidural) opioid analgesics prior to or during surgery
* Moderate to Severe pain at rest

Exclusion Criteria:

* Requires any additional surgical procedures either related or unrelated to gynecologic surgery during same hospitalization
* Procedures involving only minimal incisions such as laparotomy, laparoscopy, supraumbilical or Maylard incisions
* Has know hypersensitivity to opioids, acetaminophen, or the excipients of IV acetaminophen
* Known history of alcohol or drug abuse or misuse
* Has impaired liver function Aspartate transaminase(AST), Alanine aminotransferase(ALT), bilirubin greater than or equal to 2 times upper limit of normal
* Has significant medical disease(s), or conditions that may contraindicate participation in the study
* Has participated in another clinical trial within 30 days of surgery

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - University of Alabama (Anesthesiology), Birmingham, Alabama
  - Helen Keller Hospital, Sheffield, Alabama
  - Arizona Research Center, Inc (JC Lincoln), Phoenix, Arizona
  - Arizona Research Center, Inc. (Arrowhead), Phoenix, Arizona
  - Precision Trials, Phoenix, Arizona
  - Arcadia Methodist Hospital, Arcadia, California
  - Glendale Adventist Medical Center, Glendale, California
  - Huntington Memorial Hospital, Pasadena, California
  - Accurate Clinical Trials, Inc., San Clemente, California
  - Visions Clinical Research, Boynton Beach, Florida
  - G and G Research, Inc., Ft. Pierce, Florida
  - Century Clinical Research, INC, Holly Hill, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - University of Miami School of Medicine Dept. of Anesthesiology, Miami, Florida
  - Treasure Coast Obstetrics and Gynecology, Vero Beach, Florida
  - William Beaumont Hospital, Royal Oak, Michigan
  - Cooper Anesthesia, Camden, New Jersey
  - St. Peters University Hospital, Anesthesiology, New Brunswick, New Jersey
  - Albany Medical College Dept. of Anesthesiology, Albany, New York
  - Weill Medical College, New York, New York
  - Stony Brook Anesthesiology Health Sciences Cente, Stony Brook, New York
  - Jacobi Medical Center (Albert Einstein College of Medicine), The Bronx, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - Allegheny Pain Managment, Altoona, Pennsylvania
  - Thomas Jefferson University Dept. of Anesthesiology, Philadelphia, Pennsylvania
  - Memorial Herman/Memorial City Hospital, Houston, Texas
  - Texas Woman's Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Gynecologists and/or anesthesiologists were selected to participate as Principal Investigators.
Pre-assignment Details: Subjects were required to meet eligibility criteria prior to surgery and then again had to meet post surgical inclusion criteria.Subjects had to achieve a sufficient pain intensity score prior to entering the study.
Groups:
- IV Acetaminophen 1 g/100 mL Solution: All subjects randomized to receive Intravenous (IV) Acetaminophen 1 g/100 mL solution every 6 hours for 48 hours for a total of 8 doses.
- IV Placebo 100 mL Solution: All subjects randomized to receive Intravenous (IV) placebo 100 mL solution every 6 hours for 48 hours for a total of 8 doses.
Period: Overall Study
Arm/Group | IV Acetaminophen 1 g/100 mL Solution | IV Placebo 100 mL Solution
Started | 166 | 165
Completed | 154 | 156
Not Completed | 12 | 9
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Protocol non-compliance | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen 1 g/100 mL Solution | IV Placebo 100 mL Solution | Total
Number analyzed (Participants) | 166 | 165 | 331
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 163 | 161 | 324
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 165 | 331
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 166 | 165 | 331

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity at Rest-Baseline to 24 Hours (SPI24rest), 1 Gram IV Acetaminophen vs. Placebo.
Description: The Sum of Pain Intensity (SPI) score incorporates the analgesic effects on pain intensity (PI) from Baseline to 24 hours. SPI was measured by the 100 millimeter (mm) long Visual Analog Scale (VAS) over 24 hours after treatment. Subjects were asked to mark the level of pain they were experiencing at a certain timepoint on the scale The 100mm VAS scale was used with the left terminus (0 mm) of the scale "No Pain" and the right terminus (100 mm) with "Worst Pain Imaginable". The range of measurement is 0-2400 mm for 24 hours.
Time Frame: Baseline (just prior to the first dose) through 24 hours
Population: All efficacy analyses were conducted using the mITT population, defined as those subjects who received a complete dose of study medication prior to a request for rescue medication.
Measure: Mean (Standard Deviation); unit: units on a scale (in millimeters)
Groups:
- IV Acetaminophen 1 g/100 ml Solution: mITT Population IV acetaminophen 1 g/100 ml Solution
- IV Placebo 100 ml Solution: mITT Population IV Placebo 100 ml solution
Arm/Group | IV Acetaminophen 1 g/100 ml Solution | IV Placebo 100 ml Solution
Number analyzed (Participants) | 162 | 159
units on a scale (in millimeters) | 1793.3 (481.49) | 1845.3 (420.21)

2. Secondary Outcome: Subjects Who Experienced at Least One Treatment-emergent Adverse Event (TEAE)
Description: Number of subjects who experienced at least one treatment emergent adverse event (TEAE) A TEAE is an adverse event that occurs on or after administration of the first dose of study medication (T0)
Time Frame: First dose through 7 day follow up
Population: All analyses of safety were conducted on the Safety population, which included those subjects who received any portion of a dose of study medication.
Measure: Number; unit: Subjects
Groups:
- IV Acetaminophen 1g/100 ml Solution: Safety Population (defined as those subjects who received any portion of a dose of IV acetaminophen 1g/100 ml solution)
- IV Placebo 100 ml Solution: Safety Population(defined as those subjects who received any portion of a dose of IV Placebo 100 ml solution)
Arm/Group | IV Acetaminophen 1g/100 ml Solution | IV Placebo 100 ml Solution
Number analyzed (Participants) | 166 | 165
Subjects | 141 | 149

3. Primary Outcome: Sum Pain Intensity at Rest-Baseline to 48 Hours (SPI48rest), 1 Gram IV Acetaminophen vs. Placebo
Description: The Sum of Pain Intensity (SPI) score incorporates the analgesic effects on pain intensity (PI) from Baseline to 48 hours. SPI was measured by the 100 millimeter (mm) long Visual Analog Scale (VAS) over 48 hours after treatment. Subjects were asked to mark the level of pain they were experiencing at a certain timepoint on the scale The 100 mm VAS scale was used with the left terminus (0 mm) of the scale "No Pain" and the right terminus (100 mm) with "Worst Pain Imaginable". The range of measurement is 0-4800 mm for 48 hours.
Time Frame: Baseline (just prior to the first dose) through 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale (in millimeters)
Arm/Group | IV Acetaminophen 1 g/100 ml Solution | IV Placebo 100 ml Solution
Number analyzed (Participants) | 162 | 159
units on a scale (in millimeters) | 3612.4 (966.66) | 3718.2 (829.21)

4. Secondary Outcome: Subjects Who Experienced at Least One Treatment-emergent Serious Adverse Event.
Description: Number of subjects who reported SAEs during the study.
  A serious Adverse event (SAE) is defined as any untoward medical occurence at any dose of study medication that:
  Results in Death, Is Life Threatening, Requires inpatient hospitalization or causes prolongation of existing hospitalization, Results in persistent or significant disability/incapacity, Is a congenital anomaly/birth defect, or Is an important medical event
Time Frame: 32 days following first dose of study medication.
Measure: Number; unit: Subjects
Arm/Group | IV Acetaminophen 1 g/100 ml Solution | IV Placebo 100 ml Solution
Number analyzed (Participants) | 162 | 159
Subjects | 11 | 14

ADVERSE EVENTS:
Time Frame: Adverse Events were reported from the start of study medication until the follow up visit on Day 7 (+/- 2 days). Serious Adverse Events were collected for 32 days following start of study medication
Groups:
- IV Placebo 100 mL Solution: Safety Population (defined as those subjects who received any portion of a dose of IV Placebo 100 mL solution)
Arm/Group | IV Acetaminophen 1g/100 mL Solution | IV Placebo 100 mL Solution
Serious Adverse Events (participants affected / at risk) | 11/166 | 14/165
Other Adverse Events (participants affected / at risk) | 135/166 | 145/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Acetaminophen 1g/100 mL Solution (N=166) | IV Placebo 100 mL Solution (N=165)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 2
Vaginal infection (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 5
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aneurysm (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IV Acetaminophen 1g/100 mL Solution (N=166) | IV Placebo 100 mL Solution (N=165)
Anaemia (Blood and lymphatic system disorders) | 13 | 11
Tachycardia (Cardiac disorders) | 8 | 13
Abdominal distension (Gastrointestinal disorders) | 9 | 8
Constipation (Gastrointestinal disorders) | 48 | 49
Flatulence (Gastrointestinal disorders) | 21 | 28
Nausea (Gastrointestinal disorders) | 96 | 88
Vomiting (Gastrointestinal disorders) | 37 | 28
Pyrexia (General disorders) | 19 | 37
Dizziness (Nervous system disorders) | 10 | 16
Headache (Nervous system disorders) | 22 | 17
Insomnia (Psychiatric disorders) | 18 | 10
Pruritis (Skin and subcutaneous tissue disorders) | 24 | 21
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish only after cooperative publication or 18 months after sponsor's final evaluation of study data, whichever occurs first. At least 60 days prior to submission for publication, investigator must submit manuscript to sponsor for review and comment. Sponsor has 60 day period thereafter to respond with comment. Investigator will remove confidential information at the request of sponsor.